CLINICAL TRIAL: NCT06701409
Title: Epidemiology and Risk Factors for Injuries in Beach Tennis Players: a Prospective Cohort Study
Brief Title: Epidemiology and Risk Factors for Injuries in Beach Tennis Players
Acronym: EPITRAUMA-BT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/CHU/54; 2024-A01929-38 (Other: ANSM)
Record Dates: First submitted 2024-11-08; First posted 2024-11-22 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Sport Injury
Keywords: Beach tennis; Injuries; National prospective cohort
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Beach tennis player: After inclusion in the study, players will report their injuries monthly through an on-line questionnaire

SUMMARY:
Beach tennis, a fast-growing sport since its creation in Italy in the 1970s, has rapidly gained in popularity, particularly in La Réunion sisland since 2000. However, despite its development, studies on beach tennis-specific injuries are rare, based on cross-sectional studies and therefore limited by temporal or memory bias. The need for prospective research is crucial if we are to gain a better understanding of the epidemiology of injuries and improve prevention and medical management.

The aim will be to determine the risk of injury among beach tennis players within a one-year national prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* Player declaring that they train regularly in beach tennis (at least once a week)
* At least 18 years old at the time of inclusion
* Male or female
* Able to read and understand French
* Whether or not registered within a club
* Not opposed to the research

Exclusion Criteria:

* Protected adults (guardianship or curatorship) or those under court protection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Beach tennis players on the national territory
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Risk of injury | 1 year
  To determine the risk of injury among beach tennis players in a one-year national prospective cohort. This risk will be presented in terms of injury incidence rates.

SECONDARY OUTCOMES:
Type of injury | 1 year
  Describe the type of injury suffered by beach tennis players according to the Orchard Sports Injury Classification System (OSICS 14 classification).
Main risk factors | 1 year
  To determine the main risk factors for beach tennis injuries on the basis of variables (demographics, morphological, medical data, other sports) collected at inclusion and during follow-up.
Injury epidemiology | 1 year
  Comparing the epidemiology and characteristics of injuries between female and male players

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Bouscaren, MD, Principal Investigator — CHU de la Réunion; Julien Sebon, MD, Study Chair
Locations (1):
- CHU, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No